CLINICAL TRIAL: NCT01143454
Title: Cardiovascular Disease Discovery Protocol
Brief Title: Characterization of Patients With Uncommon Presentations and/or Uncommon Diseases Associated With the Cardiovascular System
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100126; 10-H-0126
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-10-01

CONDITIONS: Metabolic Disease; Obesity; Li-Fraumeni Syndrome; Cardiomyopathy; Atherosclerosis; Inflammatory Disease
Keywords: Cardiac Disease; iPS Cells; Cardiac Risk Factors; Cardiac Disease Discovery; Natural History; Heart Disease; Heart Disease Risk
MeSH Terms: conditions — Metabolic Diseases; Obesity; Li-Fraumeni Syndrome; Cardiomyopathies; Atherosclerosis; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1. Adult index cases and relatives: Enrolled with a known or suspected pathology that may be associated w/cardiovascular dysfunction or risk w/suspected atypical presentation, heritable disorder, or genetic predisposition.
  Interventions: Device: NSR IDE-MRI: Research pulse sequences
- 2. Child index case and child relatives: Children over 1 year of age who is affected with diseases/disorders (index cases), or who is a relative of a person who is affected with diseases/disorders.
  Interventions: Device: NSR IDE-MRI: Research pulse sequences
- 3. Healthy adult volunteers: Healthy adult volunteers must be 18 years of age or older, and must agree to have blood or tissue samples studied, and potentially stored for future research.

INTERVENTIONS:
Device: NSR IDE-MRI: Research pulse sequences — NSR IDE-MRI: Research pulse sequences, Device Manufacturer NIH. Research pulse sequences are customized pulse sequences and analysis software developed by NIH scientists.
  Groups: 1. Adult index cases and relatives; 2. Child index case and child relatives

SUMMARY:
Background:

- Researchers are interested in studying individuals who have known or suspected metabolic, inflammatory or genetic diseases that may put them at a high risk for heart diseases or diseases of their blood vessels. Depending on the condition being studied, both affected and nonaffected individuals may be asked to provide blood and other samples and may undergo tests to evaluate the heart, blood vessels and lung function. The testing is tailored to the individual and/or condition being studied. Nonaffected individuals may include relatives of affected individuals and healthy nonrelated volunteers.

Objectives:

- To study individuals who have or are at risk for cardiovascular diseases, and in some cases their unaffected relatives and healthy volunteers.

Eligibility:

- Individuals between 1 and 100 years of age. Participants may be healthy volunteers, individuals with cardiovascular diseases, or unaffected relatives of individuals with cardiovascular diseases.

Design:

* Participants will have some or all of the following tests, as directed by the study researchers:
* Photography of the face and full body
* Body measurements
* Radiography, including chest or limb x-rays
* Metabolic stress testing to study heart and muscle function
* Echocardiography to study heart function
* Magnetic resonance imaging (MRI) studies, including cardiovascular MRI, angiography, and contrast MRI, to study heart function and performance
* Computed tomography (CT) angiogram to obtain images of the heart and lungs
* Positron emission tomography (PET) imaging to study possible fat infiltration of the heart
* Six-minute walk test to study heart, lung, and muscle function and performance
* Vascular ultrasound to study blood vessel walls
* Blood, tissue, and other specimens will be collected for research and testing, and will be taken either as part of the clinical study or during surgical procedures.
* Follow-up studies may be performed under separate research protocols.

DETAILED DESCRIPTION:
We propose to characterize the etiology and natural history of rare and uncommon diseases, both known and unknown that present with symptoms and signs associated with the risk of overt or potential cardiovascular dysfunction. We will also study rare genetic modifiers and identify novel disease mechanisms contributing to common cardiovascular diseases. In so doing, we will expand our knowledge about these disorders and provide access to subjects of interest for research, teaching, and clinical experience. Individual subjects seen under this protocol may initiate the establishment of specific disease-related protocols involving intensive natural history studies, disease discovery and potential innovative therapeutic studies. In addition to its role in investigating individuals who are of interest to the Cardiovascular Branch (CB) of the NHLBI, this protocol can provide a possible avenue for admitting subjects from other NIH programs such as the NIH Undiagnosed Diseases Program, the Center for Human Immunology Trans-institute program or other NIH protocols where subjects exhibit cardiovascular features.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible subjects may include anyone over 1 year of age who is affected with diseases/disorders (index cases), or who is a relative of a person who is affected with diseases/disorders. Relatives may include genetic carriers and non-carriers.

* Healthy adult volunteers must be 18 years of age or older, and must agree to have blood or tissue samples studied, and potentially stored for future research.
* Index cases enrolled in this protocol will have been referred with a known or suspected pathology that may be associated with cardiovascular dysfunction or risk with a suspected atypical presentation, heritable disorder, or genetic predisposition. The investigator with expertise in the presentation of the subject, along with consulting specialists, will review the medical history and may review any medical records that are available of prospective subjects and offer admission based upon the potential to help the individual, to learn from the subject, or to initiate clinical or basic research suggested by the subject s workup.

EXCLUSION CRITERIA:

* Persons of less than 1 year of age or greater than 100 years of age
* Healthy volunteers unable to give informed consent or who decline to have blood and/or tissue studies, or who do not consent to have samples stored for future research may be excluded from this study.
* Pregnant women
* Persons who are not fluent in the English language will be excluded from Patient Reported Outcome Questionnaires. Such persons would be unable to properly complete questionnaires that are only valid in the English language.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Adult index cases and relatives 2. Child index case and child relatives 3. Healthy adult volunteers 4. Illiterate, Blind, or Non-English-Speaking Subjects
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-07-21 (Actual)

PRIMARY OUTCOMES:
Disease Diagnosis | Ongoing
  This protocol will allow condition-specific evaluation and sample collection to subjects with conditions associated with cardiovascular features and risk that may have long eluded diagnosis and to advance medical knowledge about rare and uncommon human diseases.

SECONDARY OUTCOMES:
Potential genetic counseling | Ongoing
  Determining molecular etiology of diseases encountered on this protocol
Understanding disease pathophysiolgy | Ongoing
  Assist in the understanding of disease pathophysiology and in the generation of diagnoses in subjects with uncommon presentations of diseases with cardiovascular consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han K, Singh K, Meadows AM, Sharma R, Hassanzadeh S, Wu J, Goss-Holmes H, Huffstutler RD, Teague HL, Mehta NN, Griffin JL, Tian R, Traba J, Sack MN. Boosting NAD preferentially blunts Th17 inflammation via arginine biosynthesis and redox control in healthy and psoriasis subjects. Cell Rep Med. 2023 Sep 19;4(9):101157. doi: 10.1016/j.xcrm.2023.101157. Epub 2023 Aug 15. PMID 37586364
- [Derived] Han K, Singh K, Rodman MJ, Hassanzadeh S, Wu K, Nguyen A, Huffstutler RD, Seifuddin F, Dagur PK, Saxena A, McCoy JP, Chen J, Biancotto A, Stagliano KER, Teague HL, Mehta NN, Pirooznia M, Sack MN. Fasting-induced FOXO4 blunts human CD4+ T helper cell responsiveness. Nat Metab. 2021 Mar;3(3):318-326. doi: 10.1038/s42255-021-00356-0. Epub 2021 Mar 15. PMID 33723462
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-H-0126.html